CLINICAL TRIAL: NCT06522906
Title: Mobilizing Hispanics With Knee Osteoarthritis Using a Dyad-based Approach: Pilot Randomized Controlled Trial
Brief Title: Mobilizing Hispanics With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Temple University (Other); University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00004081; 991639 (Other Grant/Funding Number: Rheumatology Research Foundation)
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Hispanic; Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Treatments include educational sessions about OA, a muscle strengthening program, and a program that will aim to promote regular physical activity involving dyads
  Interventions: Behavioral: Muscle Strengthening; Behavioral: General Physical Activity; Behavioral: Education
- Control (Active Comparator): Treatment only includes live video educational sessions about OA
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Muscle Strengthening — Patients will be offered five video consultations (30-45 minutes each) with a physical therapist over 3 months. The physical therapist will prescribe an exercise program individualized to the OA patient that will include strengthening exercises (2 quadriceps, 1 hip/gluteal, 1 hamstrings/gluteal, 1 calf, and 1 other) to be performed at home 3x/week.
  Arms: Intervention
Behavioral: General Physical Activity — The general program will consist of four 60-minute live video consultations conducted by a promotora. The first three sessions will be conducted every 2 weeks, with a booster session occurring one month later. The promotora will help dyads set achievable personalized physical activity goals.
  Arms: Intervention
Behavioral: Education — Administered by a promotora, treatment will include 4 live video educational sessions about OA

SUMMARY:
The objective is to conduct an early-stage clinical trial in order to provide data required to support a future clinical trial to demonstrate the effectiveness of a culturally acceptable treatment program to increase exercise and regular physical activity among Hispanics with knee osteoarthritis (OA).

Hispanic patients with knee OA paired with a chosen family member/close friend will be recruited for study participation. A pilot randomized controlled trial will be conducted. Study pairs will be randomized to receive either: 1) an intervention that will be administered by live video consultations and will include educational sessions about OA, a muscle strengthening program, and a program that will aim to promote regular physical activity involving study pairs; or 2) a control treatment that only includes live video educational sessions about OA.

Study participants will fill out a survey before the start of the study and 3 months after.

DETAILED DESCRIPTION:
Feasibility of the intervention will be based on the number of study pairs that will be recruited during the study and on attendance to the intervention sessions, and acceptability will be based on quantitative acceptability (e.g., program satisfaction) and qualitative measures.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic/Latino ethnicity
* ≥ 50 years of age
* Access to a device with internet connection
* Chronic, frequent knee pain (National Health and Nutrition Examination Survey criteria)
* Meet American College of Rheumatology criteria for knee OA WOMAC pain score of ≥4 and at least moderate pain (score 2) for at least 2 questions

Exclusion Criteria:

* Unknown or non-Hispanic ethnicity
* Condition that prevents ability to provide consent
* Illness with a life expectancy <12 months
* History of arthroplasty or prosthetic leg
* Inflammatory arthritis (e.g., rheumatoid arthritis, systemic lupus erythematosus, gout)
* Condition that prevents exercise or physical activity (e.g., unstable cardiovascular disease)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Educational sessions attended | 3 month follow-up
  Number of educational sessions attended by patients and partners will be recorded
Adherence with muscle strengthening program | 3 month follow-up
  Intervention group only. Patients will rate how much they agree/disagree (11-point numerical rating scale) with the statement: "I have been doing my exercises exactly as I was asked by my physical therapist (# sessions, exercises and repetitions)".
Adherence with physical activity plan | 3 month follow-up
  Intervention group only. Study dyads will rate how much they agree/disagree in an 11-point numerical rating scale with the statement: "I followed the physical activity plan that my promotora helped me develop".
Satisfaction with program | 3 month follow-up
  Satisfaction with the program/s, using a 7-point numerical rating scale (1="extremely unsatisfied", 7="extremely satisfied")
Perceived helpfulness | 3 month follow-up
  Perceived helpfulness of the program/s in improving OA symptoms, increasing physical activity and improving communication with their chosen partner, and the likelihood of recommending the program to OA patients and their partners, using a 5-point numerical rating scale (1=not at all/definitely would not, 5=extremely/definitely would not)

SECONDARY OUTCOMES:
Osteoarthritis disease severity | Baseline and 3 month follow-up
  Severity of OA symptoms will be measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Change in two subscale scores (joint pain [primary outcome, range 0-20] and physical function [0-68]) will be calculated.
Physical activity | Baseline and 3 month follow-up
  Physical activity will be measured using a pedometer. Participants will be asked to wear a pedometer at the waist for 7 consecutive days to record the number of steps taken per day.
Physical activity (self-report) | Baseline and 3 month follow-up
  Physical activity (self-report) of study dyads in the last week will also be measured using the Physical Activity Scale for the Elderly (range: 0-400, higher scores indicate greater physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Vina, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No